CLINICAL TRIAL: NCT02219945
Title: The Accuracy of the eNose in the Diagnostics and Monitoring of Treatment of Treatment-naive TB Patients
Brief Title: ENOSE in Pulmonary Tuberculosis in Yogyakarta
Acronym: YOGYATBNOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tjip van der Werf (Other)
Collaborators: Gadjah Mada University (Other); The Enose Company, Zutphen the Netherlands (Unknown)
Responsible Party: Sponsor-Investigator, Tjip van der Werf, Professor, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TBDIAGNOSE; KE/FK/859/EC (Registry Identifier: KE/FK/859/EC)
Record Dates: First submitted 2014-08-01; First posted 2014-08-19 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Tuberculosis Suspected; Other Specified Chronic Obstructive Pulmonary Disease; Pulmonary Tuberculosis TB (+) Histology, (-) Bacteriology
Keywords: pulmonary tuberculosis; electronic nose; diagnostic accuracy
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: 6 groups:
  1) 20 TB patients 2) 20 non-TB patients (alternative diagnosis) 3) 20 patients with chest symptoms - non-TB 4) 7 MDR-TB patients 5) 20 healthy controls 6) 300 subjects suspected to have pulmonary tuberculosis - follow-up for 2.5 years
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 - 20 PTB patients aged >18yrs (Experimental): Group 1 - 20 TB patients aged > 18 yrs 5 min exhaled breath sampling with nose clamp
  Interventions: Other: 5 min exhaled breath sampling with soft nose clamp
- Group 2 - 20 TB suspects > 18 yrs (Experimental): Group 2 - 20 non-TB patients > 18 yrs (screened for TB - but appear to test negative for TB, and diagnosed with other conditions including bronchiectasis, etc) 5 min exhaled breath sampling with nose clamp
  Interventions: Other: 5 min exhaled breath sampling with soft nose clamp
- group 3 - 20 lung patients, non-TB (Experimental): Group 3 - 20 patients with a lung disease - no TB suspects (recruited from Lung Clinics in Yogyakarta; lung cancer, COPD, etc) 5 min exhaled breath sampling with nose clamp
  Interventions: Other: 5 min exhaled breath sampling with soft nose clamp
- Group 4 - 20 healthy controls (Experimental): Group 4 - 20 apparently healthy matched controls 5 min exhaled breath sampling with nose clamp
  Interventions: Other: 5 min exhaled breath sampling with soft nose clamp
- Group 5 - 7 newly diagnosedMDR PTB pts (Experimental): Group 5 - 7 newly diagnosed MDRTB patients enrolled before start of treatment, to be followed 8 months, until after end of treatment 5 min exhaled breath sampling with nose clamp
  Interventions: Other: 5 min exhaled breath sampling with soft nose clamp
- group 6 - cohort of TB suspects (Experimental): 300 more individuals, suspected to have TB - final diagnosis by standard procedures plus sputum culture plus follow-up for >2 years 5 min exhaled breath sampling with nose clamp
  Interventions: Other: 5 min exhaled breath sampling with soft nose clamp

INTERVENTIONS:
Other: 5 min exhaled breath sampling with soft nose clamp — study participants are requested to quietly sit and allow exhaled breath to be sampled through mouth piece breathing with nose clamp during 5 min while electronic data are collected in the device and later downloaded on a laptop pc
  Other Names: AEONOSE portable exhaled breath sampling

SUMMARY:
Electronic noses detecting patterns of volatile molecules have recently been introduced for different diagnostic purposes. The diagnostic accuracy of a prototype e-nose device (Bruins et al (2013) in Bangladesh showed sensitivity of 76.5-95.9% and specificity of 85.3-98.5%. Here the investigators test a production type point-of-care hand-held device with less detectors. The investigators explore factors such as food intake, smoking, and co-morbidity, as well as the impact of TB treatment, and address the question whether the device could help monitor disease and response to treatment.

DETAILED DESCRIPTION:
Study participants provide WIC and after time for consideration, when they approve, provide demographic anonymized data.

The study population consists of six groups:

Group 1 - 20 TB patients aged > 18 yrs Group 2 - 20 non---TB patients > 18 yrs (screened for TB - other conditions) Group 3 - 20 patients with a lung disease - no TB suspects (Lung Clinics in Yogyakarta,Indonesia; Group 4 - 50 apparently healthy matched controls Group 5 - 20 newly diagnosed TB patients enrolled before start of treatment, to be followed over time, until after end of treatment (8 months FU).

Group 6 - 50 apparently healthy volunteers.

Study participants breath normally by mouthpiece into the device using a nose clamp - for 5 min during each sampling.

Electronic data are downloaded and transmitted by internet to Zutphen, Netherlands where data are processed to build the model.

ELIGIBILITY:
Inclusion Criteria:

* age >18yrs
* voluntarily participating

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
diagnostic precision of electronic nose signal in pulmonary TB | 18 months
  sensitivity and specificity of electronic nose signal in diagnosing and measuring response to treatment in pulmonary TB

SECONDARY OUTCOMES:
measuring response to TB treatment over time with the electronic nose | 18 months
  cohort of patients newly deteted with PTB will be followed with the enose device over time to monitor disease activity, until end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- patients - at 5 lung clinics (Minggiran, Kalasan, Kotagede, Bantul, Kuonprogo) connected with Sudjarto Teachnig Hospital; healthy controls among students and staff of Hospital and Gadjah Mada Universitas, Yogyakarta, Jalan Kesehatan No.1, Yogyakarta, Indonesia

REFERENCES:
- [Derived] Saktiawati AMI, Subronto YW, Stienstra Y, Sumardi, Supit F, van der Werf TS. Sensitivity and specificity of routine diagnostic work-up for tuberculosis in lung clinics in Yogyakarta, Indonesia: a cohort study. BMC Public Health. 2019 Apr 2;19(1):363. doi: 10.1186/s12889-019-6658-8. PMID 30940123